CLINICAL TRIAL: NCT01322191
Title: A Randomized Controlled Comparison of Ketorolac Tromethamine and Morphine for Postoperative Analgesia in Critically-ill, 3-18 Year-old Children: A Subgroup Analysis of Developmental Changes in Morphine Kinetics and Efficacy
Brief Title: Morphine PK Subgroup Analysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10920
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2008-03

CONDITIONS: Post Operative Pain
Keywords: pain, pain management, pediatrics, morphine pharmacokinetics
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Random assignment to a single dose of morphine 0.1 mg/kg infused by syringe pump over 10 minutes; urine and blood sample frozen at -80 degrees Celsius
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — A single dose of morphine 0.1 mg/kg infused by syringe pump over 10 minutes; urine and blood sample frozen at -80 degrees Celsius

SUMMARY:
This study was originally undertaken to evaluate the analgesic efficacy of an intravenously administered dose of ketorolac compared with intravenous morphine in the relief of acute, postoperative pain in children admitted to the Intensive Care Unit. Using the urine and plasma samples originally collected from patients in the morphine treatment group and which were never analyzed, this proposal seeks to study the pharmacokinetics and metabolism of intravenous morphine in critically-ill children along with its concentration-related efficacy using prior measures of pain.

DETAILED DESCRIPTION:
This was a randomized, double-blind, parallel, single-dose study. All children admitted to the ICU at Children's Hospital of Michigan postoperatively who required pain management were candidates. Enrollment required a Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) and/or Oucher pain score meeting the protocol definition of moderate to severe pain. Each patient was randomly assigned to receive a single dose of either morphine 0.1 mg/kg or ketorolac 0.6 mg/kg IV as the first postoperative analgesic after arriving in the ICU. Two-milliliter venous blood samples were drawn from a site contralateral to the infusion site. Samples were obtained before the dose and at 15, 30, and 60 minutes, hourly from 1-6 hours, and at 8 and 12 hours timed from the beginning of the infusion. Pain scales were assessed at the time of each pharmacokinetic sample. Plasma was immediately separated and frozen at -80°C. Urine was quantitatively collected for 12-24 hours after the study drug was administered. Urine was kept on ice at 3°C throughout the collection. At completion of the collection, the urine volume was measured and recorded, and an aliquot was frozen and maintained at -80°C. The plasma and urine samples from the morphine treated group in the original study were stored at -80°C and were not analyzed. Sets of samples of urine and plasma from 6 subjects over a range of ages have been analyzed to insure that the samples have not deteriorated during storage. This subanalysis study will provide chemical analysis of the plasma and urine samples for morphine, morphine 3 glucuronide (M3G) and morphine 6 glucuronide (M6G); pharmacokinetic analysis of morphine and its metabolites with comparison to demographics; and comparison of the morphine concentrations to the measures of analgesia. The ratio of the area under the plasma concentration vs time curves (AUC)of M6G with twice the analgesic potency as morphine and M3G with theoretical anti-analgesic properties will be compared to analgesic effects measured by the age-appropriate pain scales.

ELIGIBILITY:
Inclusion Criteria:

* All children 3-18 years of age admitted to the ICU at Children's Hospital of Michigan postoperatively who required pain management during the immediate postoperative period
* Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) and/or Oucher pain score meeting the protocol definition of moderate to severe pain

Exclusion Criteria:

* Coma (Glasgow Coma Score < 8) or significant post-operative sedation that prevented the patient from appropriate responses to questions
* Requirement of administration of a sedative or neuromuscular blocking agent, or intrathecal narcotics immediately after surgery
* Gastrointestinal hemorrhage and/or history of ulcer disease
* Frequent use of NSAIDs or narcotic analgesics for >2 weeks within the 1-month period before the study
* Asthma
* Known hypersensitivity to NSAIDs, aspirin or opiates
* Nephrotic syndrome or acute/chronic renal failure
* Thrombocytopenia (platelet count <100,000)
* Congestive heart failure
* Hepatic failure
* Treatment with methotrexate, thiazides, β-blocking agents or warfarin at the time of the study
* Dehydration or hypovolemia

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2008-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Chemical analysis of the plasma and urine samples for morphine concentration using high performance liquid chromatography coupled to atmospheric pressure ionization mass spectrometry | 2 hours

SECONDARY OUTCOMES:
Pharmacokinetic analysis of morphine, M3G, and M6G in urine to determine clearance and percent of dose excreted | 2 hours
Analgesic efficacy using drug concentration and area under the curve ratio correlated with the level of analgesia measured with the age-appropriate scale | 6 months to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ward, MD, Principal Investigator — University of Utah; Mary Lieh-Lai, MD, Principal Investigator — Children's Hospital of Michigan
Locations (2):
- United States (2):
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Utah, Salt Lake City, Utah